CLINICAL TRIAL: NCT06285526
Title: Evaluation of Perioperative Glycocalyx Monitoring in Major Abdominal Surgery
Brief Title: Glycocalyx Monitoring in Major Abdominal Surgery
Acronym: GLYCOCHIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0046/OB; 2023-A00350-45 (Registry Identifier: French Minister)
Record Dates: First submitted 2024-01-02; First posted 2024-02-29 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2023-12

CONDITIONS: Major Abdominal Surgery
Keywords: Glycocalyx; Microcirculation; Cephalic DuodenoPancreatectomy; Hyperthermic Intraperitoneal Chemotherapy
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy; Cytidine Diphosphate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group HIPEC: Cytoreduction surgery with hyperthermic intraperitoneal chemotherapy (HIPEC)
  Interventions: Procedure: Cytoreduction surgery with Hyperthermic Intraperitoneal Chemotherapy
- Group CDP: Cephalic DuodenoPancreatectomy (CDP)
  Interventions: Procedure: Cephalic DuodenoPancreatectomy

INTERVENTIONS:
Procedure: Cytoreduction surgery with Hyperthermic Intraperitoneal Chemotherapy — Cytoreduction surgery with Hyperthermic Intraperitoneal Chemotherapy
  Other Names: HIPEC
  Groups: Group HIPEC
Procedure: Cephalic DuodenoPancreatectomy — Cephalic DuodenoPancreatectomy
  Other Names: CDP
  Groups: Group CDP

SUMMARY:
The study of the microcirculation and glycocalyx could be an essential element in the monitoring of our patients undergoing major abdominal surgery. It would enable us to better target the objectives of anaesthesia and resuscitation, which until now have been based essentially on macro-circulatory parameters.

DETAILED DESCRIPTION:
This monitoring is possible in real time and real conditions by micro-camera GlycoCheck™ (Microvascular Health Solutions Inc., Salt Lake City, Utah, USA), a non-invasive monitoring allowing the study of sublingual microcirculation and glycocalyx.

ELIGIBILITY:
Inclusion Criteria:

For the HIPEC group :

* Adult patients
* Age < 75 years
* Receiving HIPEC for primary or secondary peritoneal carcinosis

For the CDP group :

* Adult patient
* Age < 75 years
* Receiving CDP for pancreatic neoplasia
* Patient who has read and understood the information letter and does not object to taking part in the study
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Secondary distant peritoneal metastases
* Chronic heart failure
* Chronic liver failure at stage C of the Child-Pugh score
* Stage IV or V chronic renal failure
* Inflammation of the sublingual buccal mucosa or injury that may locally influence sublingual microcirculation
* Patient refusal
* Person deprived of liberty by an administrative or judicial decision or person placed under court protection or guardianship

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient undergoing major abdominal surgery by cytoreduction combined with an intraperitoneal chemotherapy bath (HIPEC) or cephalic duodeno-pancreatectomy (CDP) with epidural analgesia planned in accordance with the department's usual practice
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-01-05 (Estimated); Study Completion 2025-01-05 (Estimated)

PRIMARY OUTCOMES:
Glycocalyx thickness | between the day before the operation (Day -1) and the post-operative period (Day 1)
  Perioperative variation in glycocalyx thickness (µm)

SECONDARY OUTCOMES:
Glycocalyx thickness and a biological marker of tissue hypoperfusion | post-operative period (Day 1)
  To assess, in each population ((HIPEC and CDC), the association between the thickness of the glycocalyx established by analysis of the sublingual microcirculation using GlycoCheck® and a biological marker of tissue hypoperfusion.
Glycocalyx thickness and a biological marker of tissue hypoxia | post-operative period (Day 1)
  Establish the link between glycocalyx thickness and a biological marker of tissue hypoxia.
Blood cell velocity and macrocirculatory function | post-operative period (Day 1)
  Assess the association between velocity of the red blood cells (µm/s) and cardiac index obtained by Most-Care® monitoring on Day 1.
Perfused capillary density and macrocirculatory function | post-operative period (Day 1)
  Assess the association between perfused capillary density (mm/mm2) and cardiac index obtained by Most-Care® monitoring on Day 1.
Variation of glycocalyx thickness and the daily entry-exit balance (BES) Day 1 | between Day -1 and Day 1
  To assess the difference between water and fluid intake (perfusion, nutrition, drug dilution solution) and output (diuresis, digestive aspiration, diarrhoea) over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Zoé DEMAILLY, Dr, Principal Investigator — University Rouen Hospital
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No